CLINICAL TRIAL: NCT06271122
Title: Identification of Explanatory Factors for the Lack of Muscle Strength Gain Following a Pulmonary Rehabilitation Program in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPET-1
Record Dates: First submitted 2024-01-19; First posted 2024-02-21 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Muscle weakness; Voluntary activation; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voluntary activation assessed by magnetic stimulation group (Experimental): The inclusion visit (V0) will be conducted at the beginning of the stay. On Day 1 (D+1), the patients will undergo the first visit (V1), during which specific evaluations (maximal quadriceps force test, transcranial and femoral magnetic stimulation) will be performed. Subsequently, the patients will follow the standard 4-week PR program. On Day 28 (D+28), patients will undergo the second visit (V2), during which they will undergo the same evaluations as those performed in V1.
  Interventions: Other: Voluntary activation assessed by magnetic stimulation

INTERVENTIONS:
Other: Voluntary activation assessed by magnetic stimulation — Visits V1 (Day 1) and V2 (Day 28) are identical. The dominant leg will be tested, the patient positioned on the ergometer and EMG electrodes placed on the quadriceps.
  The familiarization for femoral magnetic stimulation (FMS) will begin, the stimulation site identified and the supramaximality verified.
  After a warm up, the subject will perform 3 maximal voluntary isometric contractions (MVIC; 5s, rest = 30s), 3 MVIC reaching maximal force as quickly as possible, and 4 MVIC during which magnetic stimulation (intensity = 100%) will be applied during the contraction and 2 seconds after the contraction ends.
  For transcranial magnetic stimulation, the stimulation area and intensity will be determined. After that, the patient will perform 3 CMIV at 100%, 75%, 50% and 35% of CMIV. During each contraction, magnetic stimulation will be delivered during the force plateau.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic respiratory disease associated with various comorbidities, including muscle weakness (MW), which is very worrying due to its negative impact on patients' quality of life and survival. To address this issue, muscle strengthening is incorporated into pulmonary rehabilitation programs. However, its effectiveness is unclear, as although there is an average improvement in muscle strength, one in two patients does not show a clinically relevant improvement. To understand this non-response, it is crucial to examine the effect of muscle strengthening programs on the two main determinants of force production: the muscle and the central command. Muscle adaptations following a muscle strengthening program are well-documented, showing improvements in muscle function (cross-sectional area, lean mass, etc.). Conversely, only one study has investigated central adaptations after a muscle strengthening program, clearly demonstrating a lack of effect.

The investigators hypothesize that patients showing no improvement in muscle strength after pulmonary rehabilitation (non-responders) have a significantly lower level of voluntary activation before starting the program compared to responding patients (responders).

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic respiratory disease. Beyond respiratory symptoms, COPD is linked to comorbidities like muscle weakness (MW), significantly worrying due to its impact on patients' quality of life and survival. MW affects 32% to 57% of patients, predominantly in the lower limbs, contributing to exercise intolerance, reduced quality of life, and increased healthcare costs.

To address MW, muscle strengthening is incorporated into pulmonary rehabilitation (PR) programs. Despite significant average improvements in quadriceps muscle strength reported in the literature, a recent study highlight that 50% of patients did not clinically enhance their strength and were called non-responders (NR).

To understand this non-response, it's crucial to investigate the impact of muscle strengthening programs on the determinants of strength loss. While muscle atrophy was initially considered a major factor, studies have shown that muscle mass does not entirely explain the loss of strength. Impairment of motor control has emerged as a significant secondary determinant of muscle strength loss.

Peripheral muscle adaptations, including increased muscle surface and lean thigh mass, are well-documented. However, regarding motor control adaptations, a single study using a reference method on the quadriceps indicates a lack of effect of PR programs on central control. This observation suggests that non-responders in terms of strength may exhibit impaired motor control from the onset of the PR program.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 to 80 years
* Patients admitted to a 4-week inpatient pulmonary rehabilitation program
* Patients diagnosed with COPD (Stage I to IV) according to internationally recognized criteria determined by the GOLD
* Patients able to understanding, speaking, reading, and writing French
* Patients for whom informed consent will be obtained after a maximum 24-hour reflection period
* Patients affiliated with a French social security system or beneficiaries of such a system

Exclusion Criteria:

* Diagnosis of neurological and/or cerebrovascular disease corresponding to code 8 of the International Classification of Diseases (ICD-11)
* Possession of any invasive metallic medical devices (pacemaker, prosthesis, etc.) except for dental prostheses (crowns and bridges).
* Epileptic risk factors (chronic alcoholism, brain surgery, recent head trauma)
* Orthopedic conditions that may affect the completion of protocol tests and assessments
* Recent exacerbation (within 4 weeks)
* Patients in a period of relative exclusion compared to another protocol
* Adults protected by law or patients under guardianship or conservatorship
* Individuals deprived of liberty by a judicial or administrative decision
* Pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Central voluntary activation assessed by transcranial magnetic stimulation (TMS) | Before and after pulmonary rehabilitation (Day 1 and day 28)
  Difference in central voluntary activation (NAVcentral), representative of central command, between responders and non-responders at the beginning of a pulmonary rehabilitation program.

SECONDARY OUTCOMES:
Muscle excitability assessed by femoral magnetic stimulation (FMS) | Before and after pulmonary rehabilitation (Day 1 and day 28)
  Change in M waves's variables between responders and non-responders at the beginning and the end of the pulmonary rehabilitation program.
Contractile properties assessed by femoral magnetic stimulation (FMS) | Before and after pulmonary rehabilitation (Day 1 and day 28)
  Change in twitch's variables between responders and non-responders at the beginning and the end of the pulmonary rehabilitation program.
Corticospinal excitability assessed by transcranial magnetic stimulation (TMS) | Before and after pulmonary rehabilitation (Day 1 and day 28)
  Change in MEP's variables between responders and non-responders at the beginning and the end of the pulmonary rehabilitation program.
Intra-cortical inhibitions transcranial magnetic stimulation (TMS) | Before and after pulmonary rehabilitation (Day 1 and day 28)
  Change in MEP's silent period, representative of intra-cortical inhibitions, between responders and non-responders at the beginning and the end of the pulmonary rehabilitation program.
Voluntary activation assessed by femoral magnetic stimulation (FMS) | Before and after pulmonary rehabilitation (Day 1 and day 28)
  Change in voluntary activation (central and peripheral) between responders and non-responders at the beginning and the end of the pulmonary rehabilitation program.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Heraud, Study Director — Director of research
Locations (1):
- Clinique du Souffle La Vallonie, Lodève, France

IPD SHARING:
Plan to Share IPD: No